CLINICAL TRIAL: NCT04669301
Title: Mitigating Cancer-Related Cognitive Impairment in Older Adults With Breast Cancer Receiving Chemotherapy: Memory and Attention Adaptation Training-Geriatrics (MAAT-G): A Randomized Pilot Study
Brief Title: Memory and Attention Adaptation Training-Geriatrics (MAAT-G) Phase II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Allison Magnuson, Associate Professor - Department of Medicine , Hematology/Oncology (SMD), University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: UCCS20127; K76AG064394 (NIH)
Record Dates: First submitted 2020-12-05; First posted 2020-12-16 (Actual); Results first posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-06

CONDITIONS: Cancer-related Problem/Condition; Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Palliative Care; Time

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Supportive therapy (time and attention control) (Active Comparator): Supportive Therapy (ST) is a "behavioral placebo" and controls for non-specific psychotherapeutic factors of the clinician-subject relationship, such as empathy and support, but does not provide active cognitive training. ST utilizes reflective listening to help deepen awareness of participants' emotional experience. Timing and duration of ST sessions will mirror the intervention, and will consist of 10 weekly sessions, 30 to 45 minutes each, delivered by trained psychologists via video-conferencing.
  Interventions: Behavioral: Supportive therapy (time and attention control)
- MAAT-G intervention (Experimental): The MAAT-G intervention will be delivered by a trained psychology fellow at the University of Rochester Medical Center. The intervention will be delivered through televideoconferencing and participants will be provided a tablet equipped with a HIPPA compliant televideoconferencing application to use for the MAAT-G workshop sessions. We will use the University of Rochester Zoom application which is HIPPA compliant. A tablet instruction manual will be given to patients to help guide them through how to use a tablet and how to navigate the Zoom application. A unique meeting ID number will be given to each patient to log in to the Zoom application. If participants do not have access to wireless internet, the tablet will be equipped with a data package for participant use for the purposes of this study
  Interventions: Behavioral: MAAT-G
- Caregivers (No Intervention): Patients on this study had the option to enroll a caregiver.

INTERVENTIONS:
Behavioral: MAAT-G — Memory and Attention Adaptation Training (MAAT) is a cognitive-behavioral therapy (CBT)-based intervention for CRCD. As a CBT-based intervention, MAAT focuses on an individual's psychological response to injury as compared to the biological events triggering CRCD. MAAT is a series of manualized workshops delivered by a psychologist via video-conferencing, supplemented by a participant workbook, which provide instruction and practice with adaptive behavioral coping skills, stress management techniques, and compensation strategies.
  Arms: MAAT-G intervention
Behavioral: Supportive therapy (time and attention control) — Supportive Therapy (ST) is a "behavioral placebo" and controls for non-specific psychotherapeutic factors of the clinician-subject relationship, such as empathy and support, but does not provide active cognitive training. ST utilizes reflective listening to help deepen awareness of participants' emotional experience. Timing and duration of ST sessions will mirror the intervention, and will consist of 10 weekly sessions, 30 to 45 minutes each, delivered by trained psychologists via video-conferencing.
  Arms: Supportive therapy (time and attention control)

SUMMARY:
Cancer-related cognitive dysfunction (CRCD) affects up to 75% of patients receiving chemotherapy and older adults are at greater risk of developing CRCD, which can negatively affect their functional independence and quality of life. Memory and Attention Adaptation Training (MAAT) is a promising treatment for CRCD that improves perceived cognition in younger cancer survivors, but needs to be adapted for older adults to address their unique needs. The proposed study will adapt MAAT for older adults using feedback from key stakeholders (older adults with cancer and their caregivers), and subsequently test the ability of MAAT to improve or maintain cognition for older adults with breast cancer receiving adjuvant chemotherapy.

DETAILED DESCRIPTION:
Cancer-related cognitive dysfunction (CRCD) is a significant problem, affecting up to 75% of patients receiving chemotherapy. Older adults are at greater risk of developing CRCD which can negatively affect their functional independence and quality of life. Memory and Attention Adaptation Training (MAAT) is a promising tool that improves perceived cognition in younger cancer survivors with CRCD. For older adults with cancer, MAAT could be delivered alongside chemotherapy to mitigate the development of CRCD (when risk is highest) and CRCD-related effects on functional independence for older adults. However, MAAT will require adaptation to meet the unique needs of older adults to optimize usability and efficacy for this population. The overarching goal of this project is to adapt MAAT for older adults using input from patient and caregiver stakeholders, and subsequently gather data on the preliminary effects of the adapted MAAT (MAAT-Geriatrics [G]) on perceived cognition, objective cognitive measures and functional independence. The investigators will adapt and refine MAAT-G using feedback from key stakeholders through iterative testing of MAAT-G with 85 patient-caregiver dyads. The research plan combines the use of standardized quantitative measures of cognition and functional independence with semi-structured interviews (mixed methods), so that data from both can be integrated to optimize the adaptation and to gain a better understanding of MAAT-G's effects that are not fully captured by traditional quantitative measures alone.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of invasive breast cancer
* Planned to receive systemic therapy for breast cancer or actively receiving systemic therapy for breast cancer with two additional cycles remaining.
* Be age 65 or older
* Able to provide informed consent
* Able to read and understand English (or possess a designated health care proxy that can do the same that was designated prior to the patient losing decision-making capabilities)

Exclusion Criteria:

* Have surgery planned within 3 months of consent
* Patients who do not have decision-making capacity (decisionally or cognitively impaired) AND do NOT have a previously designated health care proxy (established prior to their cognitive impairment) available to sign consent
* Patients with breast cancer receiving endocrine therapy as their only systemic therapy will not be eligible.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 72 (Actual)
Dates: Start 2021-04-02 (Actual); Primary Completion 2024-04-17 (Actual); Study Completion 2024-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allison Magnuson, DO, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Caregivers: Patients in this study had the option to enroll a caregiver.
Period: Overall Study
Arm/Group | Supportive Therapy (Time and Attention Control) | MAAT-G Intervention | Caregivers
Started | 36 | 34 | 2
Completed | 33 | 31 | 2
Not Completed | 3 | 3 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Withdrawal by Subject | 3 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Supportive Therapy (Time and Attention Control) | MAAT-G Intervention | Caregivers | Total
Number analyzed (Participants) | 36 | 34 | 2 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 36 | 34 | 2 | 72
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 34 | 1 | 71
  Male | 0 | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 33 | 31 | 2 | 66
  Unknown or Not Reported | 3 | 2 | 0 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 2 | 0 | 6
  White | 31 | 31 | 2 | 64
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean of the Functional Assessment of Cancer Therapy-Cognition (FACT-COG)
Description: The Functional Assessment of Cancer Therapy-Cognition tool is a 50-question tool that evaluates memory and mental function in the past 7 days. The range of scores for the tool are 0 to 200 with higher scores generally indicating worse health outcomes.
Time Frame: Within four weeks of intervention completion, the intervention window was 10 weeks plus or minus 2 weeks (8 to 12 weeks).
Population: Two members of the ST population opted not to respond to the FACT-COG survey. Caregiver data was not collected for this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Supportive Therapy (Time and Attention Control) | MAAT-G Intervention | Caregivers
Number analyzed (Participants) | 34 | 34 | 0
score on a scale | 155.8 (29) | 152.7 (27.9) |

2. Secondary Outcome: Least Squares Mean for Delay Match to Sample Total Correct at the 12-second Delay (DMSTC-12) From the Cambridge Neuropsychological Test Automated Battery (CANTAB)
Description: The CANTAB Delayed Matching to Sample assesses both simultaneous visual matching ability and short-term visual recognition memory for non-verbalizable patterns. The subject is shown a complex visual pattern, followed by four similar patterns after a brief delay. The subject must select the pattern that exactly matches the sample. Better speed of response and a higher number of correct patterns indicate better health outcomes. (Patients only) The least squares mean for the variable Delay Match to Sample Total Correct at the 12-second delay (DMSTC-12) is analyzed.
Time Frame: as for outcome 1
Population: The study population missing did not have access to the technology required to complete the CANTAB, resulting in only 59 patients total rather than the 64 enrolled. CANTAB data for caregivers was not collected.
Measure: Least Squares Mean (Standard Error); unit: correct patterns
Arm/Group | Supportive Therapy (Time and Attention Control) | MAAT-G Intervention | Caregivers
Number analyzed (Participants) | 28 | 31 | 0
correct patterns | 4.04 (.17) | 4.10 (.16) |

3. Secondary Outcome: Mean of the Controlled Oral Word Association (COWA) Tool
Description: The Controlled Oral Word Association (COWA) tool is a measure of verbal fluency evaluating expressive language and executive function. Subjects are asked to freely generate as many words as they can that start with one of the prompted letters ("C", "F", and "L") in the span of one minute. Greater numbers of words indicate better health outcomes. (Patients only)
Time Frame: as for outcome 1
Population: Two members of the ST population opted not to respond to the COWA survey. Caregiver data was not collected for this measure.
Measure: Mean (Standard Deviation); unit: words generated
Arm/Group | Supportive Therapy (Time and Attention Control) | MAAT-G Intervention | Caregivers
Number analyzed (Participants) | 34 | 34 | 0
words generated | 12.4 (3.4) | 11.4 (3.2) |

4. Secondary Outcome: Mean of the Hopkins Verbal Learning Test-Revised (HVLT-R)
Description: The Hopkins Verbal Learning Test-Revised (HVLT-R) tool is a test of verbal learning and memory. Researchers read a list of 12 words to subjects and ask them to report as many of the words as they can recall. The reporting period is timed. Higher numbers of correctly remembered words, along with lower reporting times, are indicative of better health outcomes. (Patients only)
Time Frame: as for outcome 1
Population: Two members of the ST population opted not to respond to the HVLT-R survey. Caregiver data was not collected for this measure.
Measure: Mean (Standard Deviation); unit: words recalled
Arm/Group | Supportive Therapy (Time and Attention Control) | MAAT-G Intervention | Caregivers
Number analyzed (Participants) | 34 | 34 | 0
words recalled | 8 (1.8) | 7.7 (1.7) |

5. Secondary Outcome: Mean of the Geriatric Depression Screen (GDS)
Description: The Geriatric Depression Screen (GDS) tool is a 15 question psychological assessment with "yes" or "no" answers (ranging from 0 to 15, with a higher score indicating more depression). The questions pertain to emotional state and vary between positive and negative presentation. (Patients only)
Time Frame: as for outcome 1
Population: Two members of the ST population opted not to respond to the GDS survey. Caregiver data was not collected for this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Supportive Therapy (Time and Attention Control) | MAAT-G Intervention | Caregivers
Number analyzed (Participants) | 34 | 34 | 0
score on a scale | 2.3 (2.2) | 3.3 (2.4) |

6. Secondary Outcome: Mean of the Generalized Anxiety and Depression 7-item Scale (GAD-7)
Description: The Generalized Anxiety and Depression 7-item scale (GAD-7) is a 7-item question tool that evaluates feelings of anxiety over the previous 2 weeks. Each question is ranked from 0 to 3, with higher scores indicating worse health outcomes (the range for the survey is 0-21). (Patients only)
Time Frame: as for outcome 1
Population: Two members of the ST population opted not to respond to the GAD-7 survey. Caregiver data was not collected for this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Supportive Therapy (Time and Attention Control) | MAAT-G Intervention | Caregivers
Number analyzed (Participants) | 34 | 34 | 0
score on a scale | 3.4 (4.9) | 4 (4) |

7. Secondary Outcome: Mean of the Instrumental Activities of Daily Living (IADL)
Description: The Instrumental Activities of Daily Living (IADL) tool asks questions about functional independence. There are 7 questions on scale of most to least independence. The range of this scale is 3 to 21, with a higher score indicating less independence. (Patients only)
Time Frame: as for outcome 1
Population: Two members of the ST population opted not to respond to the IADL survey. Caregiver data was not collected for this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Supportive Therapy (Time and Attention Control) | MAAT-G Intervention | Caregivers
Number analyzed (Participants) | 34 | 34 | 0
score on a scale | 12.8 (2) | 12.9 (1.7) |

8. Secondary Outcome: Experience Interview - Proportion of Patients Who Expressed Perceived Benefit From Workshops.
Description: Semi-structured interview with patients about experience with workshop sessions - proportion of patients who expressed perceived benefit from workshops.
Time Frame: as for outcome 1
Population: Only 29 patients from each group (ST and MAAT-G) were selected; some patients did not allow the interview to be audiorecorded thus it was not included in the qualitative coding, thus the denominator for each group is less than in previous outcome measures. Caregiver data was not collected for this measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Supportive Therapy (Time and Attention Control) | MAAT-G Intervention | Caregivers
Number analyzed (Participants) | 29 | 29 | 0
Participants | 16 | 28 |

ADVERSE EVENTS:
Time Frame: Within four weeks of intervention completion, the intervention window was 10 weeks plus or minus 2 weeks (8 to 12 weeks).
Arm/Group | Supportive Therapy (Time and Attention Control) | MAAT-G Intervention | Caregivers
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/34 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/34 | 0/2
Other Adverse Events (participants affected / at risk) | 1/36 | 1/34 | 0/2
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Supportive Therapy (Time and Attention Control) (N=36) | MAAT-G Intervention (N=34) | Caregivers (N=2)
Memory impairment (mild) (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) — Grade 1 AE
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) — Grade 1 AE, dyspnea is discomfort when breathing
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — Grade 1 AE

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-04-02): https://cdn.clinicaltrials.gov/large-docs/01/NCT04669301/Prot_SAP_000.pdf
  • Informed Consent Form (2023-11-13): https://cdn.clinicaltrials.gov/large-docs/01/NCT04669301/ICF_001.pdf